CLINICAL TRIAL: NCT04205045
Title: Identification of Physiological Biomarkers of Gastro-intestinal Discomforts Induced by Milk Consumption
Acronym: MIDI
Status: Completed | Type: Observational
Sponsor: Paola Vitaglione (Other)
Responsible Party: Sponsor-Investigator, Paola Vitaglione, Associate Professor, Federico II University
Organization: Federico II University (Other)
Other Study IDs: MIDI
Record Dates: First submitted 2019-12-10; First posted 2019-12-19 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subjects
Keywords: milk digestibility; gastro-intestinal discomfort; milk proteins; lactose; gut permeability; gut microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, plasma pre-treated with aprotinin, urine, feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Habitual Milk Consumers (NHMC): Healthy subjects who are non-habitual milk consumers because of gastrointestinal discomforts upon milk consumption.
  Lactose breath test; Gut permeability test; Milk test.
  Interventions: Diagnostic Test: Lactose Breath Test; Other: Gut permeability test; Other: Milk Test
- Habitual Milk Consumers (HMC): Healthy subjects with regular milk consumption.
  Intervention to be performed:
  Lactose breath test; Gut permeability test; Milk test.
  Interventions: Diagnostic Test: Lactose Breath Test; Other: Gut permeability test; Other: Milk Test

INTERVENTIONS:
Diagnostic Test: Lactose Breath Test — Lactose Breath Test is performed during the recruitment step. Fasting subjects are asked to ingest 20 g of lactose in a 10% water solution. Breath samples are collected at baseline and every 30 min after lactose ingestion, for an overall test duration of 4 h. A cut-off value of 20 ppm over the baseline will be used to identify lactose malabsorbers.
Other: Gut permeability test — A 3-sugar probes test is conducted by administering 5 g lactulose, 2 g mannitol and 2 g sucralose in water solution to fasting subjects. Urine are collected at baseline (before sugar ingestion) and for time periods 0-5 h and 5-24 h.
Other: Milk Test — Milk test will be performed by administering to fasting subjects a portion of 250 ml of semi-skimmed milk treated with ultra-high temperature (UHT). Glycaemia measurements, blood withdrawals and questionnaires completion will be performed at baseline and repeated after 30 minutes, 1, 2, 4 and 6 hours after milk ingestion. Urine collection will be performed at baseline and for 6 time intervals after milk ingestion (0-2, 2-4, 4-6, 6-8, 8-12, 12-24 hours).

SUMMARY:
This study aims to explore digestibility of lactose and milk proteins, gut permeability, microbiota composition and psychological wellbeing status in healthy subjects who are non-habitual milk consumers due to milk-related gastro-intestinal discomfort in comparison with healthy and habitual milk consumers.

DETAILED DESCRIPTION:
Individuals reporting digestive disorders associated to milk and dairy products consumption increase worldwide, but in many cases this condition is not associated with a well documented diagnosis of lactose intolerance or casein allergy. Some investigators hypothesize that these disorders (in the absence of any diagnosis of disease) may be due to certain peptides forming during milk digestion. Further evidence support the hypothesis that other factors, such as a lacking activity of intestinal brush border enzymes, an altered gut permeability, and/or a specific gut microbiota composition, may be involved in the onset of gastrointestinal (GI) discomforts induced by milk consumption. Indeed, all these factors could modulate the amount and type of peptides and lactose skipping digestion and passing through the intestinal mucosa, leading to effects on GI motility and gastro-intestinal hormone secretion. Similarly, due to its implications in homeostatic and non-homeostatic regulation of eating behaviour as well as in pain-regulating processes, a role of endocannabinoid system (ECs) in the evolution of GI symptoms post-milk consumption could be hypothesized.

In this study, the digestibility of lactose and milk proteins will be explored in healthy subjects who are non-habitual milk consumers (NHMC) because of gastro-intestinal discomforts induced by milk ingestion, in comparison with healthy and habitual milk consumers (HMC). The gut permeability, the composition of intestinal microbiota and the psychological wellbeing status of subjects will be also investigated and compared in the 2 groups.

The study design, after the enrollment of participants based on pre-recruitment questionnaires and a lactose breath test, includes a gut permeability test and a milk test.

The potential eligibility of subjects to participate in this study will be assessed through pre-recruitment questionnaires, collecting personal and socio-demographic data of volunteers, information about milk consumption habits and associated symptoms, general information about health (anthropometry, health status, smoking and alcohol consumption habits), household environment, information on volunteer's consideration about milk product and its consumption, and food habits.

Potential eligible subjects who will sign the informed consent form, will be assessed for final eligibility by mean of a lactose breath test, performed according to the protocol approved during the Rome Consensus Conference (2009). GI symptoms will be also recorded by subjects, in parallel with H2 measurements in breath samples and up to 24 hours from the beginning of the test, by mean of Visual Analogue Scales (VAS).

During the lactose breath test, subjects will be asked to fill out the physical activity questionnaire (short version of the IPAQ), questionnaires on quality of life, on depression, anxiety and stress (DASS), a semi-quantitative food frequency questionnaire (FFQ), the King's Stool Chart, to evaluate frequency and consistency of feces, and the Three Factor Eating Questionnaire (TFEQ) to evaluate individual eating behaviour. Anthropometric data of weight and height will be measured as well.

The overall symptoms evolved during and after the lactose breath test will be assessed together with the H2 concentrations measured in breath samples; a cut-off value of 20 ppm over the baseline will be used to identify lactose malabsorbers.

This selection procedure will identify as eligible:

* subjects who are negative to breath test (BT-) and do not refer any GI symptom (lactose absorber) or refer some minor gastro-intestinal symptoms
* subjects who are positive to breath test (BT+) but without any symptom (lactose malabsorbers without symptoms).

On the other hand, subjects will be excluded from the study if:

* they are positive to breath test (BT+) and report GI symptoms (lactose intolerant)
* they are negative to breath test (BT-) but report severe GI symptoms such as "vomiting" and "Loose, mushy or watery stools".

The enrollment will be concluded when 2 groups of subjects will be constituted as follow

* Group 1, habitual milk consumers (HMC): 20 subjects who are regular milk consumers (>700 mL/week), do not experience GI discomfort after milk intake and are lactose tolerant or lactose malabsorber.
* Group 2, non-habitual milk consumers (NHMC): 20 subjects who are not regular milk consumers (< 150 mL/week), because of GI discomforts after milk intake and are lactose tolerant or lactose malabsorber.

For all subjects from both groups the gut permeability test and the milk test will be performed. These tests will be scheduled after one week from the lactose breath test and with one week in between. Subjects will be also asked to collect a fecal sample under usual dietary habits.

For gut permeability test, subjects will receive instruction about drug consumption and will be asked to follow a controlled diet for 2 days before the test (avoiding milk and dairy products, and food products containing polyols).

Fasting subjects will collect a baseline urine sample, before drinking a solution containing 5 g lactulose, 2 g mannitol and 2 g sucralose in 100 ml of water. Urines will be collected for time periods 0-5 h and 5-24 h in two containers added with 1 mL of a chlorhexidine solution at 1 ppm. Urine samples collected over 24 h and delivered the day after to the study centre will be aliquoted (1.5 ml) and frozen at -20°C until analyses.

During the week before the milk test, subjects will fill a food diary. Moreover they will be instructed to not drink any milk, dairy product and any food product containing milk proteins during the 2 days before the milk test. On the day of milk test, fasting subjects will fill out questionnaires about their actual appetite and GI symptoms, baseline urine and blood samples will be collected, and fasting glycaemia by finger-prick will be measured. Subsequently, subjects will drink 250 ml of milk within 10 min and thereafter, glycaemia, symptoms and appetite questionnaires, as well as blood samples and urine will be collected at specific time points. After the last blood drawing subjects will be offered a lunch and, before leaving the study centre, they will be instructed to fill out GI symptoms and appetite questionnaires, to collect urine, to fill out a food diary, and to consume a fixed dinner. Questionnaires, diaries and 6-24h urine samples will be delivered to the laboratory on the next day.

Blood samples, stored at -40°C will be analyzed for:

* gastro-intestinal hormones (insulin, gastric inhibitory peptide (GIP), glucagon-like peptide 1 (GLP-1), glucagon, c-peptide, ghrelin, leptin) in plasma samples pre-treated with aprotinin;
* endocannabinoids and N-acyl-ethanolamines (ECs);
* casein digestion-derived peptides (beta-casomorphins and all known peptides derived from milk proteins);
* aminoacid profile;
* DPPIV activity;
* baseline DPPIV concentration.

Urine samples, aliquoted (1.5 ml) and frozen at -40°C, will be used to measure:

* lactose, galactose + glucose, and indican excretion levels (for urines collected over 24 h after milk test).
* lactulose, mannitol and sucralose excretion levels (for urines collected over 24 h after gut permeability test).

Fecal samples, stored at -40°C, will be used for DNA extraction according to the standard operating procedures of the International Human Microbiome Consortium (http://www.human-microbiome.org/). Statistical analysis will be carried out by the most appropriate methods in order to infer the associations between specific microbiota signatures and clinical, dietary and metabolomic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Drinking milk (maximum 150 ml/week for non-habitual milk consumers and minimum of 700 ml/week for habitual milk consumers)
* BMI between 18.5 - 30 kg/m2
* Available for three visits (with one week in between).
* Willing to drink 250 ml of milk in fasting condition within 10 min
* Written informed consent
* Negative lactose breath test result (increase in H2 concentrations < 20 ppm vs basal value) and without symptoms or with any symptoms except "vomiting" and "Loose, mushy or watery stools"
* Lactose malabsorbers (increase in H2 concentrations > 20 ppm vs basal value but without symptoms)

Exclusion Criteria:

* Presence of any relevant organic, systemic or metabolic disease or abnormal laboratory values.
* Ascertained intestinal organic diseases, including celiac disease or inflammatory bowel diseases.
* Previous major abdominal surgeries.
* Active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment are also acceptable).
* Untreated food intolerance.
* Lactose intolerant
* Assumption of probiotics or topic and/or systemic antibiotic therapy during the last month.
* Systematical/frequent assumption of contact laxatives.
* Pregnant and lactating women.
* Inability to conform with protocol.
* Treatment with any investigational drug within the previous 30 days.
* Recent history or suspicion of alcohol abuse or drug addiction.
* Subjects having symptoms of "vomiting" and "Loose, mushy or watery stools" at any level of severity following milk consumption and the lactose breath test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample. Recruitment will be done through public announcements in the department places, local ambulatories and shops, and invitation through social networks.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in plasmatic concentration of milk-derived peptides following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of casein digestion-derived peptides (beta-casomorphins and all known peptides derived from milk proteins) in plasma samples by mean of HPLC-MS/MS.
Changes from baseline of insulin plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of insulin by mean of Luminex kits in plasma samples pre-treated with aprotinin.
Changes from baseline of glucose-dependent insulinotropic peptide (GIP) plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of GIP by mean of Luminex kits in plasma samples pre-treated with aprotinin.
Changes from baseline of glucagon-like peptide 1 (GLP-1) plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of GLP-1 by mean of Luminex kits in plasma samples pre-treated with aprotinin.
Changes from baseline of glucagon plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of glucagon by mean of Luminex kits in plasma samples pre-treated with aprotinin
Changes from baseline of c-peptide plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of c-peptide by mean of Luminex kits in plasma samples pre-treated with aprotinin.
Changes from baseline of ghrelin plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of ghrelin by mean of Luminex kits in plasma samples pre-treated with aprotinin.
Changes from baseline of leptin plasmatic levels following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of leptin by mean of Luminex kits in plasma samples pre-treated with aprotinin.
Changes from baseline in serum levels of endocannabinoids and N-acyl-ethanolamines response following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of endocannabinoids N-acyl-ethanolamines in serum by mean of HPLC-MS/MS
Increases from baseline in urinary concentration of lactose following milk ingestion. | baseline and time intervals (0-2, 2-4, 4-6, 6-8, 8-12 and 12-24 hours) following milk ingestion.
  Measure of lactose and galactose + glucose excreted in urine samples by mean of high pressure liquid chromatography coupled with tandem mass spectrometry (HPLC-MS/MS).

SECONDARY OUTCOMES:
Changes from baseline in plasmatic concentration of milk-derived aminoacids following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of aminoacids in plasma samples by mean of HPLC-MS/MS.
Changes from baseline of glycaemia following milk ingestion. | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  Measure of glycaemia by finger pricking and using a bedside glucometer.
Changes from baseline in gastro-intestinal symptoms developed after milk ingestion. | Baseline and at 0.5, 1, 2, 4, 6, 8, 12 and 24 hours after milk ingestion.
  Evaluation of gastro-intestinal symptoms occurrence and intensity with Visual Analog Scale (Area Under the Curve) over time for each symptoms
Concentration of baseline serum DPPIV | baseline
  DPPIV' s concentration in serum samples by mean of immuno-enzymatic assay with Luminex kit.
Activity of serum DPPIV | baseline and at 0.5, 1, 2, 4 and 6 hours after milk ingestion.
  DPPIV' s activity in serum samples by mean of spectrophotometric assay.
Changes from baseline in urinary concentration of indican over 24 h following milk ingestion | baseline and time intervals (0-6 and 6-24 hours) after milk ingestion.
  Measure of indican by mean of HPLC-MS/MS as marker of protein digestibility.
Association of GI symptoms with appetite, glycaemia, plasmatic GI hormones and milk-derived peptides/aminoacids over the first 6 hours post milk consumption, as well as with urinary lactose and galactose + glucose over 24 hours post milk consumption. | Baseline and 0.5, 1, 2, 4, 6 hours post milk ingestion for blood biomarkers, and at baseline and time intervals (0-2, 2-4, 4-6, 6-8, 8-12, 12-24 hours) post milk ingestion for analytes in urines.
  Association will be evaluated by mean of statistical analyses including correlation and regression analysis.
Increases from baseline in urinary concentration of lactulose, mannitol and sucralose over 24 h after oral challenge as markers of intestinal permeability. | baseline and time intervals (0-5 and 5-24 hours) after oral challenge.
  Measure of lactulose, mannitol and sucralose by mean of HPLC-MS/MS. Lactulose/Mannitol (L/M) ratio in the urine collected within 5 hours after oral challenge represents the small intestinal permeability; the total amount of sucralose in the 24 h urine represents the colonic permeability.
Gut microbiota composition | One sample
  Faecal samples must be collected by subjects under habitual dietary conditions (without any restriction about milk/milk-derived products and at least 4 days after the gut permeability test). Microbiota composition will be determined by high throughput sequencing of the 16S ribosomal ribonucleic acid (rRNA) gene. The massive number of sequences obtained will be analyzed by using state of the art bioinformatics tools and the presence and relative abundance of the microbial species occurring in each sample will be determined.
Prevalence of lactose malabsorption in the two groups (assessed with Lactose Breath Test). | During recruitment step
  Measure of H2 levels in breath samples collected before (in fasting condition) and after oral administration of 20 g of lactose. A cut-off value of 20 ppm over the baseline will be used to identify lactose malabsorbers.
psychological profile | During recruitment step
  evaluation of psychological wellbeing of subjects for each group by mean of questionnaires about perception of quality of life, depression, anxiety and stress, and eating behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vitaglione, PhD, Study Director — Federico II University
Locations (1):
- Department of Agricultural Sciences, Portici, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We will decide as soon as we will have data analysis completed and a clear idea on publication rute according with the other coauthors.

REFERENCES:
- [Derived] Tagliamonte S, Puhlmann ML, De Filippis F, Guerville M, Ercolini D, Vitaglione P. Relationships between diet and gut microbiome in an Italian and Dutch cohort: does the dietary protein to fiber ratio play a role? Eur J Nutr. 2024 Apr;63(3):741-750. doi: 10.1007/s00394-023-03308-4. Epub 2023 Dec 27. PMID 38151533

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT04205045/Prot_SAP_002.pdf